CLINICAL TRIAL: NCT02386462
Title: To Determine the Median Effective Dose (ED50) of Dexmedetomidine to Facilitate LMA Insertion During Anaesthesia Induction With Propofol 2.0 mg/kg
Brief Title: Determine the ED50 of Dexmedetomidine to Facilitate LMA Insertion During Anaesthesia Induction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Guangzhou General Hospital of Guangzhou Military Command (Other)
Responsible Party: Principal Investigator, bo xu, associate chief physician, Guangzhou General Hospital of Guangzhou Military Command
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LMA insertion
Record Dates: First submitted 2015-03-06; First posted 2015-03-12 (Estimated); Last update posted 2015-03-12 (Estimated); Status verified 2014-12

CONDITIONS: Anesthesia
Keywords: laryngeal mask airway; circulatory reflexes
MeSH Terms: interventions — Dexmedetomidine; Propofol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dexmedetomidine (Experimental): After an injection of pre-determined bolus dose of dexmedetomidine over 10 min, anaesthesia was induced with propofol 2.0 mg/kg. The modified Dixon's up-and-down method was used to determine the bolus dose of dexmedetomidine, starting from 1.0μg/kg (step size; 0.1μg/kg).
  Interventions: Drug: Dexmedetomidine; Drug: Propofol

INTERVENTIONS:
Drug: Dexmedetomidine — The modified Dixon's up-and-down method was used to determine the bolus dose of dexmedetomidine, starting from 1.0μg/kg (step size; 0.1μg/kg)
Drug: Propofol

SUMMARY:
Dexmedetomidine can be used as a co-induction agent to facilitate laryngeal mask airway (LMA) insertion with minimal effect on respiratory function. The purpose of the study was to determine the median effective dose (ED50) of dexmedetomidine to facilitate LMA insertion during anaesthesia induction with propofol 2.0 mg/kg.

DETAILED DESCRIPTION:
Dexmedetomidine is a highly selective α2 receptor agonist, which produces sedative, anxiolytic and analgesic effects without causing clinically significant respiratory depression. Dexmedetomidine also reduces the propofol requirement for sedation and anaesthesia induction. Therefore, dexmedetomidine may be a useful co-induction agent to facilitate LMA insertion with minimal effects on respiratory function. A recent study showed that dexmedetomidine administration prior to propofol induction provided similar conditions for successful LMA insertion, as does fentanyl without respiratory depression. The purpose of this study was to determine the median effective dose (ED50) of dexmedetomidine required for successful LMA insertion during induction with propofol of 2 mg/kg .

ELIGIBILITY:
Inclusion Criteria:

1. ASA Ⅰ ~ Ⅱ women undergoing Laparoscopic surgery.
2. Written informed consent from the patient or the relatives of the participating patient.
3. BMI:18.5～25

Exclusion Criteria:

1. Mental illness can not match
2. epidural anesthesia contraindicated
3. People who have Slow-type arrhythmias
4. Chronic renal failure
5. Alcohol or drug abuse
6. Already taking gabapentin, pregabalin, benzodiazepin or antidepression drug

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-11; Primary Completion 2015-04 (Estimated); Study Completion 2015-04 (Estimated)

PRIMARY OUTCOMES:
The assessment of sedation (determine the effect-site dose of dexmedetomidine blunting cardiovascular responses to the insertion of the laryngeal mask airway at the same level of sedation) | 5min after the end of the infusion
  The aim of this study was to determine the effect-site dose of dexmedetomidine blunting cardiovascular responses to the insertion of the laryngeal mask airway at the same level of sedation.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Military Region General Hospital, Department of Anesthesiology, Guangzhou, Guangdong, China